CLINICAL TRIAL: NCT06419712
Title: Effect of Vitamin D Supplementation on Glutathione Peroxidase (GPx) Activity, Interleukin-6 (IL-6) Levels and Clinical Outcomes in Post-COVID-19 Patients
Acronym: VITDPOSTCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escuela Militar de Graduados de Sanidad, SEDENA (Other)
Responsible Party: Principal Investigator, IVÁN IGNACIO MEJÍA, DR. IVÁN IGNACIO MEJÍA, Escuela Militar de Graduados de Sanidad, SEDENA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C32-22
Record Dates: First submitted 2024-05-15; First posted 2024-05-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Post-COVID19 Condition
Keywords: Post-COVID-19 condition; long-COVID-19; vitamin D; cholecalciferol; interleukin-6; glutathione peroxidase; cough; dyspnea; fatigue; anxiety; depression
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Cough; Dyspnea; Fatigue; Anxiety Disorders; Depression | interventions — Vitamin D; Cholecalciferol; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily Vitamin D Supplementation Group (Experimental): This arm of the study involves daily administration of vitamin D to participants, with the dosage adjusted based on body weight and initial vitamin D levels, aiming to achieve and maintain optimal serum vitamin D levels
  Interventions: Drug: vitamin D (cholecalciferol) supplementation
- Weekly Bolus Vitamin D Supplementation Group (Experimental): This arm of the study involves administering a weekly bolus dose of vitamin D, equivalent to the total daily dose accumulated over the week, to investigate the efficacy of this regimen in improving vitamin D levels and reducing post-COVID-19 symptoms.
  Interventions: Drug: vitamin D (cholecalciferol) supplementation

INTERVENTIONS:
Drug: vitamin D (cholecalciferol) supplementation — This clinical pilot study administered and compared daily and bolus dosing regi-mens of vitamin D to achieve and maintain optimal serum levels of 25(OH)D in post-COVID patients. The daily dose group received constant and gradual supplementation of cholecalciferol, intended to achieve more stable 25(OH)D levels without peaks. Conversely, the bolus group received a weekly dose that could lead to rapid increases followed by gradual declines in 25(OH)D levels. The Daily dose of cholecalciferol was calculated using the following formula: Daily dose of cholecalciferol = [Weight (kg) × desired increase in 25(OH)D (ng/ml) × 2.5] - 10 .

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of vitamin D supplementation in treating neuropsychiatric symptoms and improving antioxidant levels in individuals diagnosed with post-COVID-19 condition, a state known as long-COVID. These individuals are primarily adults who have recovered from severe COVID-19 and exhibit persistent symptoms. The main questions it aims to answer are:

Does vitamin D (cholecalciferol) supplementation decrease levels of anxiety and depression in patients with post-COVID-19 condition? Does vitamin D (cholecalciferol) supplementation increase glutathione peroxidase (GPx) activity in these patients? Researchers will compare the effects of daily versus bolus doses of vitamin D (cholecalciferol) to see if one method is more effective than the other in achieving sufficient vitamin D levels and improving clinical outcomes.

Participants will:

Be randomly assigned to receive either a daily dose or a bolus dose of vitamin D over an 8-week period.

Undergo blood tests to measure biochemical markers such as interleukin-6 (IL-6) and GPx before and two months after starting supplementation.

Have their lung function tested using spirometry and diffusing capacity for carbon monoxide.

Complete the Hospital Anxiety and Depression Scale to assess changes in anxiety and depression levels.

DETAILED DESCRIPTION:
This clinical trial investigates the potential therapeutic benefits of vitamin D supplementation in individuals experiencing persistent health issues following recovery from severe COVID-19, commonly referred to as post-COVID-19 condition or long-COVID. The study primarily focuses on the neuropsychiatric symptoms such as anxiety and depression and the antioxidant enzyme activity, specifically glutathione peroxidase (GPx), which plays a critical role in mitigating oxidative stress within the body.

The trial is designed as a pilot, randomized controlled trial, where participants are divided into two groups to receive vitamin D in different dosing regimens: a daily dose and a bolus dose, administered weekly. This method allows for an examination of the efficacy of dosage frequency on achieving optimal serum vitamin D levels, which are hypothesized to influence the biochemical pathways involved in inflammatory and oxidative processes.

During the study, participants' serum levels of 25-hydroxyvitamin D (25(OH)D), a marker for vitamin D status, are assessed to ensure they reach and maintain a target level that previous studies have associated with optimal immune function and reduced inflammation. The participants' initial vitamin D status is carefully evaluated to tailor the supplementation dose according to individual needs, following a formula that considers their weight and the desired increase in 25(OH)D levels.

The antioxidant capacity of participants is measured through the activity of GPx in the blood. This enzyme is crucial for reducing oxidative stress, which is linked to various chronic diseases and has been suggested to play a significant role in the severity and progression of post-COVID-19 symptoms. By measuring GPx activity before and after vitamin D supplementation, the study aims to provide insights into the effectiveness of vitamin D in enhancing antioxidant defenses in post-COVID patients.

Furthermore, the trial includes an evaluation of lung function using high-resolution computed tomography (HRCT) and standard pulmonary function tests, including spirometry and the diffusing capacity of the lung for carbon monoxide (DLCO). These assessments help to determine any improvements in respiratory health, which is often compromised in patients with long-term COVID-19 effects.

The impact of vitamin D on neuropsychiatric symptoms is assessed using the Hospital Anxiety and Depression Scale (HADS), a validated tool that rates the severity of anxiety and depression symptoms. This aspect of the study highlights the potential of vitamin D not just as a physical health supplement but also as a modulator of mental health, particularly in the context of the ongoing recovery from a severe infectious disease.

By conducting this trial, the researchers aim to shed light on the broader implications of vitamin D supplementation, not only as a means of improving vitamin D status but also as a potentially significant intervention for improving the quality of life and health outcomes in individuals suffering from long-term effects of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Post-COVID-19 Condition: Patients must have been previously diagnosed with COVID-19 and continue to experience persistent symptoms after recovery.
* Age: Participants must be adults aged 18 years or older.
* Vitamin D Deficiency: Initial serum 25-hydroxyvitamin D levels below 40 ng/mL.
* Completed Hospital Treatment for COVID-19: Patients must have been discharged from hospital treatment for COVID-19 at least 12 months prior to the study.
* Ability to Give Informed Consent: Participants must be capable of understanding and willing to sign a consent form.
* Ability to Perform Required Tests: Participants must be physically able to undergo spirometry and other functional tests as required by the study protocol.

Exclusion Criteria:

* Reading and Writing Difficulties: Patients who have difficulties in reading and/or writing that would impede their understanding of the study requirements or communication with study staff.
* Inability to Perform Physical Tests: Patients unable to perform functional walk and spirometry tests.
* Untreated Chronic Non-Respiratory Diseases: Individuals suffering from untreated chronic diseases such as diabetes mellitus, systemic arterial hypertension, hypothyroidism, or epilepsy that could interfere with the study outcomes.
* Recent Use of Vitamin D Supplements: Patients who have taken vitamin D supplements within three months prior to the start of the study.
* Participation in Other Clinical Trials: Patients currently participating in other clinical trials that might conflict with this study's protocol.
* Pregnancy: Due to potential risks and lack of data on high-dose vitamin D supplementation during pregnancy, pregnant women will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Glutathione Peroxidase (GPx) Activity | Baseline and two months post-supplementation
  This measure assesses the antioxidant enzyme activity level in the blood, indicating the body's capacity to reduce oxidative stress. Increased activity of GPx is expected as a result of vitamin D supplementation
Serum Levels of Interleukin-6 (IL-6) | Baseline and two months post-supplementation.
  IL-6 is a pro-inflammatory cytokine. The study aims to observe changes in IL-6 levels, which might not be significantly altered by vitamin D supplementation as per preliminary findings.

SECONDARY OUTCOMES:
Lung Function Tests | Baseline and two months post-supplementation.
  Includes Forced Vital Capacity (FVC) and Forced Expiratory Volume in One Second (FEV1). Improvements in these parameters would suggest beneficial effects of vitamin D on lung health
Neuropsychiatric Symptoms (Anxiety and Depression) | Baseline and two months post-supplementation.
  The severity of anxiety and depression will be quantified using the Hospital Anxiety and Depression Scale (HADS). A decrease in HADS scores post-supplementation is anticipated.

OTHER OUTCOMES:
Symptoms of Cough, Dyspnea, and Fatigue | Baseline and two months post-supplementation.
  Assessment of respiratory and general symptoms associated with long-COVID to determine any subjective improvement post-vitamin D supplementation
Serum 25-Hydroxyvitamin D Levels | Baseline and two months post-supplementation.
  This measure will confirm the efficacy of the vitamin D supplementation regimen in achieving and maintaining sufficient serum levels of vitamin D.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, and after publication of the primary findings, the following Individual Participant Data will be made available:
  Anonymized Participant Data: This includes all individual data collected during the trial, minus any personally identifiable information. Data types include:
  Demographic information (age, gender, etc.) Clinical data (symptoms, disease severity, etc.) Treatment data (dosage received, treatment duration, etc.) Outcome data (response to treatment, side effects, etc.) Laboratory results (vitamin D levels, IL-6 levels, GPx activity, etc.).